CLINICAL TRIAL: NCT05003427
Title: 68Ga-FAPI-04 PET/CT for the Detection of Oral Carcinoma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCH-OralFAP
Record Dates: First submitted 2021-08-06; First posted 2021-08-12 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Oral Carcinoma
Keywords: PET/CT; FAPI
MeSH Terms: conditions — Mouth Neoplasms | interventions — 68Ga-FAPI

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-FAPI-04 PET/CT (Experimental): The patients were injected with 55.5-148 MBq (1.5-4mCi) of 68Ga-FAPI-04 in one dose intravenously and underwent SPECT/CT scan 30-90 min later.
  Interventions: Drug: 68Ga-FAPI-04

INTERVENTIONS:
Drug: 68Ga-FAPI-04 — 68Ga-FAPI-04 were injected into the patients before the PET/CT scans

SUMMARY:
FAPI is a fibroblast activation protein inhibitor and 68Ga-FAPI-04 is a potential new imaging agent for imaging of carcinoma. 68Ga-FAPI-04 PET/CT is helpful to clarify the benign, malignant and invasive range of the oral carcinoma, locate and qualitatively diagnose the tumor, and make early diagnosis and restaging of recurrent tumor.

DETAILED DESCRIPTION:
Sometimes, the traditional 18F-FDG PET/CT diagnosis of head and neck tumors mistakenly diagnosed inflammatory lymph nodes as metastatic lymph nodes, resulting in false positive results. Fibroblast activation protein (FAP) is a serine peptidase on the surface of tumor associated fibroblasts. It plays an important role in promoting the growth, invasion, metastasis and immunosuppression of tumor cells. FAPI is a fibroblast activation protein inhibitor and 68Ga-FAPI-04 is a potential new imaging agent for imaging of carcinoma. 68Ga-FAPI-04 PET/CT is helpful to clarify the benign, malignant and invasive range of the oral carcinoma, locate and qualitatively diagnose the tumor, and make early diagnosis and restaging of recurrent tumor.

ELIGIBILITY:
Inclusion Criteria:

* patients in suspicion of oral carcinoma,
* 68Ga-FAPI-04 and 18F-FDG PET/CT within 2 week;
* being able to provide basic information and sign the written informed consent form.

Exclusion Criteria:

* claustrophobia,
* pregnancy,
* breastfeeding,
* kidney or liver failure,
* inability to fulfill the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance1 | 1 year
  comparing the SUV and number of Oral cancer or metastasis detected by 68Ga-FAPI-04 and 18F-FDG PET/CT
Diagnostic performance2 | 1 year
  comparing the SUV and number of Oral cancer or metastasis detected by 68Ga-FAPI-04 and 18F-FDG PET/CT

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Science and Peking Union Medical College, Beijing, Beijing Municipality, China